CLINICAL TRIAL: NCT00514059
Title: Open Clinical Study to Assess the Immune Response and Safety of a Booster Dose (5th Dose) of a Combination Vaccine Against Diphteria-Tetanus-Pertussis-Polio Given to Healthy Adolescents 15-16 Years of Age.
Brief Title: Immunogenicity and Safety Study of a Booster Dose (5th) of Diphteria-Tetanus-Pertussis-Polio Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SM07-01
Record Dates: First submitted 2007-08-08; First posted 2007-08-09 (Estimated); Last update posted 2007-08-09 (Estimated); Status verified 2007-04

CONDITIONS: Diphtheria; Tetanus; Pertussis; Polio
Keywords: Diphteria-tetanus-pertussis-polio vaccine; Booster immunization; Vaccine effect (Diphtheria-tetanus-acellular pertussis-polio); Immunity; Safety
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough; Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Drug: Boostrix polio

INTERVENTIONS:
Drug: Boostrix polio — 1 dose (0.5 ml) i.m.

SUMMARY:
An open clinical trial to study the immune response and safety after giving a booster dose (5th Dose) of a combination vaccine against Diphteria-Tetanus-Pertussis-Polio to healthy adolescents 15-16 Years of age. The first three doses were given during the first year of life, according to the Norwegian child immunization program. The fourth dose was given in a previous clinical trial performed in 1998 when the children were 6-7 years old.

In 2006 there was a change in the child immunization program in Norway: a fourth dose of a Combination Vaccine Against Diphteria-Tetanus-Pertussis-Polio is given to children 6-7 years old.

This study will give us information if there is need for an additional dose (5th dose) of a combination vaccine, containing the pertussis components, before the adolescents are leaving secondary school.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adolescents who have previously received a dose of a vaccine against diphteria, tetanus, pertussis and polio in a clinical trial in 1998
* Written informed consent from the adolescent and one of his/her parents
* The family must understand norwegian

Exclusion Criteria:

* Serious chronic diseases
* Vaccination against tetanus last 12 months
* Immunization with a Diphteria vaccine component after the study in 1998
* Suspected or confirmed immune deficiency
* Immunological/immunosuppressive treatment
* Pregnancy
* Serious reactions to previous immunization with any of the vaccine components
* Acute fever (axillary temperature ≥ 38°C) at the the of vaccination. (Postpone vaccination)

Ages: 15 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2007-04; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
To measure vaccine specific antibody responses after a fifth dose of a combination vaccine against diphteria-tetanus-pertussis-polio. To register local and systemic reactions after vaccination.

SECONDARY OUTCOMES:
To measure vaccine specific antibody responses approximately eight years after a fourth dose of a combination vaccine against diphteria-tetanus-pertussis-polio.

CONTACTS AND LOCATIONS:
Overall Officials: Synne Sandbu, Physician, Principal Investigator — Norwegian Institute of Public Health
Locations (1):
- Norwegian Institute of Public Health, Oslo, Norway